CLINICAL TRIAL: NCT03942783
Title: A Randomised Controlled Trial of Job Retention Vocational Rehabilitation for Employed People With Inflammatory Arthritis: the WORKWELL Trial.
Brief Title: WORKWELL: Testing Work Advice for People With Arthritis
Acronym: WORKWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Collaborators: University of Central Lancashire (Other); University of Manchester (Other); Versus Arthritis (Other)
Responsible Party: Principal Investigator, Yeliz Prior, Professor Yeliz Prior, University of Salford
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UoSWORKWELL1.1
Record Dates: First submitted 2018-09-08; First posted 2019-05-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Arthritis, Inflammatory
Keywords: work rehabilitation; vocational rehabilitation; occupational therapy; rehabilitation; presenteeism; employment
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Arthritis | interventions — Rehabilitation, Vocational

STUDY DESIGN:
Intervention Model Description: The WORKWELL trial is a definitive, pragmatic, patient-blinded, multi-centre superiority randomised parallel group trial of: a) WORKWELL compared to b) written work self-help advice in people with RA, UIA or PsA. Both groups will continue to receive usual care. The primary endpoint is the summed score of the Work Limitations Questionnaire-25 (a measure of work presenteeism) at 12 months after baseline assessment.
  2022 update: An extension to the study had been approved to complete a 36 month follow-up.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigators will remain blinded to group allocation until the participant has completed and returned their baseline questionnaire, and the data verified at the Lancashire CTU.
  Data co-ordination staff at the CTU, who will be responsible for contacting patients to obtain missing data from 6- and 12-month questionnaires will be blinded to group allocation. The Data Manager and Information Systems team will be unblinded.
  Due to the nature of the intervention it will not be possible for therapists to be blinded to group allocation. Participants cannot be blinded to the intervention they receive.
  The statistician will be blinded to group allocation by using a dummy variable for group allocation until analysis is complete. The health economist will not be blinded as the costs of WORKWELL will need to be included into the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The control group will receive a written work self-help information pack plus usual care. The pack includes published arthritis patient information booklets about work; a decision-tree flowchart; information about the UK Equality Act. The self-help information pack is mailed to the participants by the CTU following randomisation.
  Usual care consists of: prescribed medication; attending Rheumatology clinics; referral to rehabilitation, as and when deemed necessary from the Rheumatology clinic, but not including work advice. Any rehabilitation required will be provided as normal, e.g. provision of exercise, self-management education, activities of daily living advice, psychosocial support.
  Interventions: Other: Control
- WORKWELL Group (Experimental): The same as the Control Group (i.e. self-help information pack, plus usual care) PLUS the WORKWELL intervention. This consists of, on average, 4.5 hours contact, including: a structured work assessment; identification of work-related barriers and priority problems; collaborative treatment planning with the participant; a range of self-management, work advice and job modifications appropriate to the individual participant's problems; goal setting and action planning; and a 30 minute telephone review to identify progress with goals at the end of treatment.
  Interventions: Other: WORKWELL

INTERVENTIONS:
Other: WORKWELL — Individualised, tailored work advice and work/vocational rehabilitation, including self-management and job modifications.
  Other Names: Vocational rehabilitation; Work rehabilitation
  Arms: WORKWELL Group
Other: Control — Published arthritis work booklets;written guidance on work problem identification; potential actions
  Other Names: written work self-help information pack
  Arms: Control Group

SUMMARY:
Background: Inflammatory arthritis (IA) causes work disability, absenteeism (sick leave) and presenteeism (reduced productivity) at high cost to individuals, employers and society. A trial of job retention vocational rehabilitation (VR) amongst people with IA in the US showed that VR reduced work disability. However, it is unknown whether this approach transfers to the United Kingdom (UK) with a different social and welfare structure. Previously, we modified the VR for the UK, funded by Arthritis Research UK (the WORKWELL programme) and demonstrated it to be deliverable and acceptable in a feasibility trial. Our aim now is to move to the definitive UK trial testing the effectiveness and cost-effectiveness of WORKWELL.

Methods: A multicentre randomized controlled trial will be conducted. Employed people with rheumatoid, psoriatic or inflammatory arthritis (n=240), with concerns about continuing working due to arthritis, will be randomized to receive WORKWELL or control (written advice). WORKWELL includes individualised VR (maximum 4.5 hours over several months): assessing work problems; encouraging arthritis self-management in the workplace; addressing ergonomics; considering fatigue and stress management; providing orthoses and educating on employment rights and support services, assistive technology and work modifications. It also includes psychological and disclosure support, workplace visits and employer liaison (as applicable). Outcomes will be assessed at 0, 6 and 12 months by questionnaire. The primary outcome is the Work Limitations Questionnaire-25 (measuring presenteeism: summed score) at 12 and 36 months, with cost-effectiveness analysis at 12 months.

Discussion: If effective and cost-effective, WORKWELL can be rolled out in Rheumatology services to help improve the quality and duration of people with arthritis' working lives.

DETAILED DESCRIPTION:
Background Work problems are common in people with inflammatory arthritis (IA). In rheumatoid arthritis (RA) 33% stop working within two years and 50% within 10 years. Work difficulties include: pain (particularly hand pain); fatigue; unadapted work environments, equipment and work schedules; poor work self-efficacy (i.e. lack of confidence about working); job strain; limited use of self-management strategies; and limited support from employers and work colleagues. Two USA trials of brief (3 hours) job retention vocational rehabilitation (VR) identified job loss was postponed by modifying such factors. A UK proof-of-principle trial (n=32) identified 10 hours (minimum) of VR reduced work instability. VR is not routinely available in the NHS and Rheumatology departments. It is unclear from the evidence if brief VR provided by therapists is effective and cost-effective in the UK.

Aims

1. Assess if there is a difference in work presenteeism between people with RA, undifferentiated IA (UIA) or psoriatic arthritis (PsA) who receive either: usual care, written work self-help information plus brief VR (WORKWELL) provided by a therapist trained in providing VR; or usual care and written work self-help information only (WP1).
2. To assess if there are differences in self-reported work instability, work, activity limitations, work productivity, absenteeism, work status, work self-efficacy, health status, NHS and societal costs between people receiving WORKWELL or written work self-help information only (WP1)
3. To assess the cost-effectiveness of WORKWELL from the perspective of: the NHS using health-related quality of life as the primary outcome; the employer using presenteeism as the primary outcome; and the employer using health-related quality of life as the primary outcome and including presenteeism as a cost. (WP5)
4. To update and evaluate a VR programme for occupational therapists and physiotherapists to help them keep people with RA, IA or PsA in work (WP2).
5. To measure fidelity to the WORKWELL intervention (WP3).
6. To understand the social and structural context in which the intervention is delivered and to identify factors which may influence the quality of implementation (WP3).
7. Investigate contextual factors influencing participants' presenteeism (WP4).

Design A pragmatic, multi-centre individually randomised controlled trial (RCT) comparing the effects of brief VR (intervention) with written self-help advice only (control). Cost-effectiveness and process evaluations will also be conducted.

Methodology Employed people with RA/ UIA/ PsA who have concerns about being able to continue to work in future due to arthritis, will be consented into the study. They will complete a baseline questionnaire (hard copy or online according to participant preference) and will then be randomly allocated in equal numbers, stratified by participants' job skill levels, to either intervention or control groups. Participants (in both groups) will be mailed a self-help work information pack. Participants' in the intervention group will be referred to receive the WORKWELL intervention from a trained occupational therapist/ physiotherapist. The Lancashire Clinical Trials Unit (CTU: University of Central Lancashire) will contact participants monthly by text/ e-mail/ telephone to identify numbers of days on sick leave. Six months after completing the baseline questionnaire, participants will complete a short postal/online questionnaire including presenteeism, productivity health status measures and resource data. At 12 months, participants will complete a third postal/online questionnaire with most of the measures collected at baseline. Two sub-samples from the intervention and control groups will be interviewed: employed participants about their views of VR; and any unemployed/ retired due to ill-health participants about factors contributing to job loss. At 36 months, participants will complete a fourth postal/online questionnaire with some of the key work status measures collected at baseline. Two sub-samples from the intervention and control groups will be interviewed: employed participants about their views of VR; and any unemployed/ retired due to ill-health participants about factors contributing to job loss.

Planned Sample Size 240 people will be recruited from 18 sites. On completion of the trial, qualitative interviews will be completed with 15 employed participants and up to 7 (if any) unemployed / early retired through ill-health from the intervention group. WORKWELL participants' line managers/employers will also be interviewed (where possible: n=10). WORKWELL Therapists and their line managers will also be interviewed (one each from each site, or less if data saturation is reached (n=18 for each).

Analyses Statistical analyses will investigate differences in outcomes at 12 and 36 months after baseline between intervention and control groups using mixed effects linear, logistic or ordinal logistic regression modelling, adjusted for baseline values and stratification variables (as applicable). The primary outcome is the summed score of the Combined Work Activities Limitations Scale -Work Limitations Questionnaire-25 (a measure of work presenteeism) at 12 and 36 months after baseline assessment. The health economic analysis will be conducted from the UK National Health Service (NHS) and employer perspectives. Interviews will be thematically analysed. Records will be analysed using content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (i.e. aged ≥ 18 years)
* diagnosed with RA, UIA or PsA by a Rheumatology Consultant. (Undifferentiated Inflammatory Arthritis is defined as: persistent synovitis in more than one small joint of the hand, without any other known cause, but the person does not yet meet all the diagnostic criteria for RA. Participants can have co-morbidities (which may also be related to having RA, UIA or PsA, for example, osteoarthritis, fibromyalgia, heart condition, mild to moderate anxiety or depression; or are unrelated, e.g. diabetes.
* In paid work (full or part-time, self-employed or contractual work) for at least 15 hours per week.
* Participants may be on sick leave at the time of screening BUT this must be for less than 4 weeks duration and not planned or likely to extend for longer than 4 weeks.
* Able to read and understand English.
* Score ≥10 on the RA-Work Instability Scale (RA-WIS), a measure of mismatch between the person's abilities and their job demands.
* Able to attend the participating site for WORKWELL appointments, if allocated to that group
* Able to provide informed consent.

Exclusion Criteria:

* on extended sick leave (i.e. > 4 weeks). The WORKWELL intervention is designed for people currently in work. Long-term sick leave is defined as being > 4 weeks [NICE, 2009b].
* Already planning to retire due to age or to take early retirement (for any health or non-health reason) within the next 12 months (i.e. within the trial follow-up period)
* planning to move out of area within the next 3 months and therefore would be unable to attend for WORKWELL sessions if allocated to that group (as treatment may not be completed in time).
* already receiving or awaiting VR services from Access to Work or a Vocational Rehabilitation company. These services conduct work assessments as part of VR provision. (Those receiving work services from other sources (e.g. occupational health or human resources in their organisation, online advice from Fit for Work) may still be recruited as VR provision can be of varied quality and this will be considered as "usual care."
* Employed in the armed forces (as they could be stationed overseas during the trial period. The armed services also have their own Vocational Rehabilitation service.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Combined Work Activities Limitations Scale - Work Limitations Questionnaire-25 | Change between 0 to 12 months; 0 to 36 months
  Measure of presenteeism (i.e. productivity at work). Scale range 0-111Higher values indicate worse outcome

SECONDARY OUTCOMES:
Rheumatoid Arthritis Work Instability Scale | Change 0 to 12 months
  Measure of the degree of mismatch between functional abilities and workplace demands. Scale range 0-23. Higher scores indicate worse problems.
Work status | Change between 0 and 12 months; 0 to 36 months
  Options are whether in full- or part-time work; early retired; retired; unemployed
Absenteeism | Monthly for 12 months
  Number of days sick leave/month. Total number of sick days over 12 month period is calculated.
Work Self-Efficacy Scale | Change 0 to 12 months
  Confidence about working; 0-10 scale; higher scores indicate greater confidence
Work Productivity and Activity Impairment Scale | Change 0 to 12 months
  Measures time off on sick leave or for any other reason, hours worked; health problems effect on work productivity and ability to do other daily activities; percentage absenteeism - all in the last 7 days.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as follows:
  Scoring instructions available at: http://www.reillyassociates.net/WPAI_Scoring.html
Short Form-12 (SF-12) Health Survey | Change 0 to 12 months
  Physical and mental health.
EuroQol Five Dimensions QuestionnaireEQ5DL-5 | Change 0 to 12 months.
  Quality of Life Scale
Rheumatoid Arthritis Impact of Disease Scale | Change 0 to 12 months
  Domains of impact of RA: coping, helplessness, fatigue, physical function, sleep, global assessment and pain.
  RAID final value = (pain NRS value (range 0-10) x 0.21) + (function NRS value (range 0-10) x 0.16) + (fatigue NRS value (range 0-10) x 0.15) + (phys well being NRS value (range 010) x 0.12) + (sleep NRS value (range 0-10) x 0.12) + (emotional well being NRS value (range 0-10) x 0.12) + (coping NRS value (range 0-10) x 0.12).
  Thus, the range of the final RAID value is 0-10 where higher figures indicate worse status.
RA Disease Activity Index-5 | Change 0 to 12 months
  The RADAI contains five items on global disease activity during the past 6 months (item 1), current disease activity as measured by swollen and tender joints (item 2), current amount of arthritis pain (item 3), current duration of morning stiffness (item 4) and current number of tender joints in a joint list (item 5). The first three items are scored on an 11-point numerical rating scale, with verbal anchors from ''no disease activity''/''no pain'' (score 0) to ''extreme disease activity''/''extreme pain'' (score 10). The last two items are scored on a seven-point (item 4) and four-point (item 5) verbal rating scale.
Health Resource Use Questionnaire | cumulative health recourse use over 12 months
  Measure of health resource use (secondary and primary care; social care; private health care)

OTHER OUTCOMES:
The Perceived Workplace Support Scale | Change 0 to 12 months
  Perceived level of managerial, co-worker and organisational support available to respondent. Each subscale is scored by adding the scores. Sub-scale a: managerial support score range 4 to 20; co-worker support scale b range 8-40; organisational support scale c score range 7-35. Higher scores indicate less support
The Work Transitions Index | Change 0 to 12 months;
  Work disruptions due to arthritis
Work-Health - Personal Life Perceptions Scale: short form | Change 0 to 12 months
  Ability to balance demands of work, health and personal life. Score range 4 - 16, higher score indicates worse balance
The Workplace Accommodations, Benefits, Policies and Practices Scale | Change 0 to 12 months
  a) The number of job accommodations, policies and workplace practices employees have available in their workplace (range 0 - 17), and b) how helpful they find it helpful each of these to manage health related work difficulties (1 to 5 scale). Higher scores indicate greater level of helpfulness

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Prior, PhD, Principal Investigator — University of Salford
Locations (18):
- United Kingdom (18):
  - North Bristol NHS Trust, Bristol, Avon
  - Countess of Chester Hospital NHS Foundation Trust, Chester, Cheshire
  - Newcastle Upon Tyne Hospitals NHS Trust., Newcastle upon Tyne, Co Tyne and Wear
  - Northern Devon Healthcare NHS Trust, Barnstaple, Devon
  - NHS Fife, Kirkcaldy, Fife
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - St Helens and Knowsley Teaching Hospitals NHS Trust, St Helens, Merseyside
  - Aneurin Bevan University Health Board, Chepstow, Monmouthshire
  - Northumbria Healthcare NHS Foundation Trust, Hexham, Northumberland
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - The Royal Wolverhampton NHS Trust, Cannock, Staffordshire
  - Cardiff and Vale UHB: LLandough Hospital, Cardiff, Vale of Glamorgan
  - Royal United Hospitals Bath NHS Foundation Trust, Bath, Wiltshire
  - Worcestershire Acute Hospitals NHS Trust, Worcester, Worcestershire
  - Barnsley Hospitals NHS Foundation Trust, Barnsley, Yorkshire
  - The Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
UK Work Environment Survey (work assessment: already open access). Workwell Solutions Manual to be shared at end of trial (open access).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At end of trial.
Access Criteria: Application to study team

REFERENCES:
- [Background] Battista S, Parker J, Ching A, Culley J, Long S, Heard A, Hammond A, Radford K, Holland P, O'Neill T, Walker-Bone K, Prior Y. WORKWELL process evaluation: qualitative data analyses of the participant interviews at 12- and 36-month follow-ups. Rheumatol Adv Pract. 2025 Mar 14;9(2):rkaf034. doi: 10.1093/rap/rkaf034. eCollection 2025. PMID 40124973
- [Background] Hammond A, Sutton C, Cotterill S, Woodbridge S, O'Brien R, Radford K, Forshaw D, Verstappen S, Jones C, Marsden A, Eden M, Prior Y, Culley J, Holland P, Walker-Bone K, Hough Y, O'Neill TW, Ching A, Parker J. The effect on work presenteeism of job retention vocational rehabilitation compared to a written self-help work advice pack for employed people with inflammatory arthritis: protocol for a multi-centre randomised controlled trial (the WORKWELL trial). BMC Musculoskelet Disord. 2020 Sep 10;21(1):607. doi: 10.1186/s12891-020-03619-1. PMID 32912199
- [Background] Sutton C, Cotterill S, Forshaw D, Rhodes S, Haig A, Hammond A. SWAT 86 evaluation: Randomised evaluation of prenotification of trial participants before self-report outcome data collection to improve retention. Research Methods in Medicine and Health Sciences 2022 3(4): 107-115 https://doi.org/10.1177/26320843221098427
- [Background] Hammond A, Radford KA, Ching A, Prior Y, O'Brien R, Woodbridge S, Culley J, Parker J, Holland P. The Workwell trial: protocol for the process evaluation of a randomised controlled trial of job retention vocational rehabilitation for employed people with inflammatory arthritis. Trials. 2022 Nov 9;23(1):937. doi: 10.1186/s13063-022-06871-z. PMID 36352479
- [Background] Ching A, Parker J, Haig A, Sutton CJ, Cotterill S, Forshaw D, Culley J, Hammond A. Job retention vocational rehabilitation for employed people with inflammatory arthritis: adaptations to the WORKWELL trial due to the impact of the COVID-19 pandemic. Trials. 2022 Dec 20;23(1):1030. doi: 10.1186/s13063-022-06941-2. PMID 36539794
- [Derived] Hammond A, O'Brien R, Woodbridge S, Prior Y, Ching A, Culley J, Parker J. Upskilling Rheumatology Occupational Therapists in Work Rehabilitation: An Evaluation of a Job Retention Vocational Rehabilitation Training Course (the Workwell Trial). Musculoskeletal Care. 2025 Mar;23(1):e70067. doi: 10.1002/msc.70067. PMID 40022440
- [Derived] Hammond A, O'Brien R, Woodbridge S, Parker J, Ching A. The Work Experience Survey - Rheumatic conditions (United Kingdom): Psychometric properties and identifying the workplace barriers of employed people with inflammatory arthritis receiving vocational rehabilitation. Musculoskeletal Care. 2023 Dec;21(4):1578-1591. doi: 10.1002/msc.1835. Epub 2023 Oct 25. PMID 37876334